CLINICAL TRIAL: NCT03158805
Title: A Randomized, Placebo-Controlled Study of Liraglutide 3mg Daily (Saxenda®) in Obese or Overweight Patients With Stable Bipolar Disorder
Brief Title: Saxenda® in Obese or Overweight Patients With Stable Bipolar Disorder (Investigator Initiated)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Lindner Center of HOPE (Other)
Responsible Party: Principal Investigator, Susan McElroy, Chief Research Officer, Lindner Center of HOPE
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2017-1579
Record Dates: First submitted 2017-05-15; First posted 2017-05-18 (Actual); Results first posted 2024-03-27 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-03

CONDITIONS: Bipolar Disorder; Obesity
MeSH Terms: conditions — Bipolar Disorder; Obesity | interventions — Liraglutide

STUDY DESIGN:
Intervention Model Description: We will conduct a single-center, randomized, placebo-controlled, double-blind, parallel-group, 2-arm clinical trial of liraglutide 3.0 mg sc injection in 60 obese or overweight outpatients with stable BP.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Active drug (Active Comparator): LIRAGLUTIDE 3 Mg/0.5 mL (18 Mg/3 mL) SUB-Q PEN INJECTOR (ML)
  Interventions: Drug: LIRAGLUTIDE
- Placebo (Placebo Comparator): Placebo (no active drug)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: LIRAGLUTIDE — 3 Mg/0.5 mL (18 Mg/3 mL) SUB-Q PEN INJECTOR (ML)
  Other Names: Saxenda
  Arms: Active drug
Other: Placebo — Placebo injection
  Arms: Placebo

SUMMARY:
Taken together these data support the hypothesis that liraglutide 3.0 mg sc injection will reduce body weight and improve metabolic variables in obese or overweight patients with BP without worsening psychiatric symptoms. The investigators predict that liraglutide 3.0 mg sc injection will display greater efficacy as compared to placebo in decreasing body weight in patients with BP who are obese or overweight. To prove this hypothesis, investigators will conduct a single-center, randomized, placebo-controlled, double-blind, parallel-group, 2-arm clinical trial of liraglutide 3.0 mg sc injection in 60 obese or overweight outpatients with stable BP. The investigators have chosen BP rather than another SMI because it is the most common SMI (more common than schizophrenia or schizoaffective disorder) and has a particularly strong association with obesity.

DETAILED DESCRIPTION:
BACKGROUND AND SIGNIFICANCE:

Obesity is common among persons with severe mental illness (SMI), especially those with bipolar disorder (BP) (1-5). It is estimated that 45-55% of people with SMI are obese, making obesity 1.5-2 times more common among those with SMI than among the general population. Indeed, in a recent pragmatic lithium trial conducted in BP, 69% of the subjects were overweight or obese. Although the precise mechanism underlying the relationship between obesity and SMI is unknown, it is thought to be multifactorial, involving genetic factors, intrinsic features of SMI (e.g., overeating, poor dietary choices, sedentary lifestyle, and sleep dysregulation), and the weight-gaining effects of most of the psychotropic medication used to treat SMI.

Importantly, obesity is thought to contribute to the well-documented elevated mortality from cardiovascular disease (CVD) among those with BP. Thus, weight reduction in obese people with BP might be important for reducing their morbidity and mortality from CVD and other obesity-related conditions (e.g., diabetes and metabolic syndrome). Conversely, the presence of obesity in patients with BP is associated with a more severe course of illness , a lower health-related quality of life (18), reductions in brain gray and white volumes (19, 20), and non-adherence with antipsychotic medications . Indeed, it has been hypothesized that successful treatment of obesity in those with BP might benefit mental as well as physical health. It is thus imperative that obesity be a focus of treatment in those with BP.

Comprehensive behavioral weight management programs have shown some effectiveness for obesity in patients with SMI, but the weight loss is modest at best and such programs are difficult to implement and not widely available. Several medications have been shown to mitigate psychotropic-induced weight gain, particularly metformin and topiramate, but many patients either do not respond to these agents or are unable to tolerate them. Importantly, the efficacy and safety of newly available weight-loss agents have not been evaluated in people with SMI.

In December 2014, the U.S. Food and Drug Administration approved liraglutide [rDNA origin] 3 mg/day subcutaneous [sc] injection) (Saxenda®) as a treatment option for chronic weight management in individuals with obesity. The drug is approved for use in adults with a body mass index (BMI) of 30 or greater (obesity) or adults with a BMI of 27 or greater (overweight) who have at least one weight-related comorbid condition such as hypertension, type 2 diabetes, or dyslipidemia, in combination with reduced-calorie diet and increased physical activity. Liraglutide is a glucagon-like peptide-1 (GLP-1) receptor agonist. Saxenda® and Victoza® contain the same active ingredient (liraglutide) at different doses (3 mg and 1.8 mg, respectively). However, unlike Victoza®, Saxenda® is not indicated for the treatment of type 2 diabetes, as the safety and efficacy of Saxenda® for the treatment of diabetes has not been established.

Several lines of evidence suggest that liraglutide 3.0 mg sc injection (Saxenda®), in combination with a reduced-calorie diet and increased physical activity, would be a useful weight-loss treatment for patients with BP who are overweight or obese.

First, GLP-1 is a gut/brain peptide that is secreted from intestinal mucosal enteroendocrine L cells in response and in proportion to nutrient stimulation of the gut, and that suppresses food intake by acting on receptors in key areas of the brain that regulate energy balance (e.g., hypothalamus and hindbrain) (34-37). In humans, administration of GLP-1 reduces food intake and increases satiation in a dose-dependent manner (37). Obesity in people with BP, as well as psychotropic-induced weight gain, are thought to be due to in part to increased food intake (2). It is thus possible that liraglutide 3.0 mg sc injection will decrease food intake in obese patients with BP, thereby reducing body weight.

Second, preliminary preclinical and clinical findings suggest liraglutide 3.0 mg sc injection may be effective for antipsychotic-induced weight gain and antipsychotic-induced obesity (38). Thus, liraglutide has been shown to produce weight loss in animal models of olanzapine-induced weight gain. In one of these studies, liraglutide also produced antidepressant-like effects. (Indeed, other animal studies suggest that liraglutide may have antipsychotic properties. In the only published case of liraglutide use in a patient with SMI, an obese (BMI 33.5=mg/kg2) 60-year-old woman with schizophrenia treated with clozapine, liraglutide (1.8mg/day) produced a sustained weight loss of 7.7 kg (an 8.7% body weight reduction) over two years. Liraglutide was well tolerated and there were no psychiatric adverse events (i.e., the patient's schizophrenia remained stable). At our own center, we have treated a 32-year-old woman with schizoaffective disorder, bipolar type and obesity (BMI=36 mg/kg2) receiving one depot and two oral antipsychotics with liraglutide 3.0 mg sc injection and, to date, she has lost 7.5 kg (an 8.3% body weight reduction) over a 4-month period. She reports the liraglutide 3.0 mg sc injection has reduced her hunger and improved her satiety. She has tolerated liraglutide 3.0 mg sc injection well and has had no difficulties with giving herself the injections, her psychological symptoms have remained stable, and there have been no adverse psychiatric effects. Indeed, her mild tardive dyskinesia is much improved

Third, relative to other weight loss agents, liraglutide 3.0 mg sc injection has a favorable psychiatric and cardiovascular adverse event profile. Regarding psychiatric events, in the pivotal liraglutide 3.0 mg sc injection clinical trials, 6 (0.2%) of 3384 liraglutide 3.0 mg sc injection-treated patients had suicidal ideation (one of these individuals made a suicide attempt) compared with none of the 1941 placebo-treated patients. Additionally, 2.4% of liraglutide 3.0 mg sc injection recipients had insomnia and 2.0% had anxiety, compared with 1.7% and 1.6 %, respectively, of placebo recipients. Conversely, lorcaserin (Belviq®) was associated with euphoria (0.2% vs < 0.1% for placebo) and is contraindicated in patient's receiving serotonergic medications (and many psychotropics enhance serotonin function). Phenermine/topiramate combination (Qsymia®), at the highest approved dose, was associated with insomnia (11.1% vs 5.8% for placebo), depression/mood problems (7.6% vs 3.4% for placebo), and anxiety (7.9% vs 2.6% for placebo). Additionally, one of the components of Qsymia®, topiramate, is associated with suicidality. Bupropion/naltrexone combination (Contrave®), at the highest recommended dose, was associated insomnia (9.2% vs 5.9% for placebo), anxiety (4.2% vs 2.8% for placebo), and irritability (2.6% vs 1.8% for placebo). Moreover, there are reports of components of these latter medications (e.g., phentermine and bupropion) causing severe adverse psychiatric events, such as mania and psychosis. Taken together, these findings suggest that liraglutide 3.0 mg sc injection may be the least likely of these weight management medications to exacerbate psychiatric symptoms in people with BP. Indeed, GLP-1 analogues have been reported to produce enhanced well-being in patients with diabetes.

Taken together these data support the hypothesis that liraglutide 3.0 mg sc injection will reduce body weight and improve metabolic variables in obese or overweight patients with BP without worsening psychiatric symptoms. We predict that liraglutide 3.0 mg sc injection will display greater efficacy as compared to placebo in decreasing body weight in patients with BP who are obese or overweight. To prove this hypothesis, we will conduct a single-center, randomized, placebo-controlled, double-blind, parallel-group, 2-arm clinical trial of liraglutide 3.0 mg sc injection in 60 obese or overweight outpatients with stable BP. We have chosen BP rather than another SMI because it is the most common SMI (more common than schizophrenia or schizoaffective disorder) and has a particularly strong association with obesity.

RESEARCH DESIGN AND METHODS

Study hypothesis (es):

The central research question is whether liraglutide 3.0 mg sc injection is efficacious for reducing body weight in obese or overweight patients with BP. We hypothesize that liraglutide 3.0 mg sc injection will be an efficacious, safe, and well tolerated treatment for weight loss in obese or overweight patients with stable BP. We predict that liraglutide 3.0 mg sc injection will display greater efficacy as compared to placebo in decreasing body weight in patients with BP who are overweight or obese without increasing psychiatric adverse events. We also predict that liraglutide 3.0 mg sc injection will produce a greater percentage of patients who lose ≥ 5% of baseline body weight, and improve BMI, waist circumference, fasting lipid and glucose levels, HgA1c levels, and measures of eating psychopathology.

Endpoints:

The primary endpoint will be the percent change in body weight from Baseline (Week 0) to week 40/Early Termination (ET) (see Table 1 for a schedule of assessments). Secondary endpoints will include proportion of participants who lose ≥ 5% of baseline body weight, and change from baseline in body weight (kg), BMI, waist circumference, and metabolic variables (fasting lipids and glucose, and HgA1c levels). Exploratory secondary endpoints will be change from baseline in eating psychopathology, assessed with the Three Factor Eating Questionnaire (TFEQ) and Binge Eating Scale (BES). Safety endpoints assessed at each study visit will be mental status examination, clinically-administered scales that assess psychopathology (CGI-BP scale [both Severity and Improvement subscales], YMRS, MADRS, and CSSRS), vital signs, and adverse events determined by clinical interview. Laboratory tests and 12-lead electrocardiograms (ECGs) will be obtained at Screening, week 8, week 16/ET, and week 40/ET. Compliance will be assessed at each visit with inspection of returned multi-dose pens. Potential interactions between liraglutide and psychiatric medications will be monitored and recorded on the Potential Drug Interaction form (see p. 28).

Study type:

This is a single-center, randomized, placebo-controlled, double-blind, two-arm, parallel-group, fixed-dose efficacy and safety study with 3 phases: a 3-27 day Screening period; a 40-week randomized, double-blind Treatment period (4 weeks of dose titration and 36 weeks of dose maintenance); and a 1-week Follow-up (drug discontinuation) period. The purpose of the 40-week Blinded Treatment phase is to establish the efficacy of liraglutide 3.0 mg sc injection for weight loss in obese patients with stable BP.

Study population:

We expect to screen about 90 subjects in order to randomize 60 subjects in a 1:1 ratio to drug or placebo. Patients will be recruited from the Lindner Center of HOPE, Mason, OH, a University of Cincinnati College of Medicine Affiliate. Patients will be recruited by clinician referral and advertisement.

Participants will include 60 outpatients with a DSM-5 diagnosis of BP that is stable, who are obese or overweight with at least one weight-related comorbidity, and who have been receiving a stable psychotropic regimen for the past three months. The weight-related comorbidities to be included will be hypertension, type 2 diabetes, and dyslipidemia. Allowed psychotropic medications for BP will include mood stabilizers (lithium, valproate, and lamotrigine), antipsychotics (asenapine, aripiprazole, cariprazine, chlorpromazine, clozapine, haloperidol, loxapine, olanzapine, paliperidone, perphenazine, quetiapine, resperidone, thiothixene, trifluoperazine, or ziprasidone), antidepressants, and anxiolytics (benzodiazepines, gabapentin or pregabalin, and buspirone). Stable BP will be operationally defined as a CGI-BP-Severity score of 1through 3 (1= normal, not at all; 2= borderline mentally ill; 3=mildly ill); a YMRS score ≤12; a MADRS score ≤19, and the absence of clinically significant suicidality and psychosis. Participants must be 18 through 65 years of age, be able to provide informed consent, and if female, be postmenopausal, surgically incapable of childbearing, or practicing a medically acceptable method(s) of contraception (e.g., hormonal method, intrauterine device) for at least 1 month prior to study entry and throughout the study. Exclusion criteria include subjects with a lifetime DSM-5 Axis I diagnosis of dementia, a psychotic or depressive disorder, or a substance use disorder within the past three months; those with clinically significant psychotic features or suicidal ideation; those with serious or unstable general medical illnesses; those with a personal or family history of medullary thyroid cancer or Multiple Endocrine Neoplasia syndrome type 2; those who are allergic to or who have demonstrated hypersensitivity to liraglutide 3.0 mg sc injection or any of its components; and females who are pregnant, nursing, or intend to become pregnant. Specific entry criteria are listed below.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women, ages of 18-65 years, inclusive.
2. Participants will have a DSM-5 bipolar disorder that is clinically stable.
3. Participants will have received a stable major psychotropic drug regimen (except for minor dosage adjustments) for at least 3 months prior study entry. Major psychotropic drugs are antipsychotics, mood stabilizers, and antidepressants. Subjects may have had changes in adjunctive benzodiazepines and hypnotic agents.
4. Participants will be obese (defined as a BMI ≥ 30 mg/kg2) or overweight (defined as BMI ≥ 27 kg/m2) with at least one weight-related comorbidity, such as hypertension, type 2 diabetes, or dyslipidemia.

5 Participants in treatment for a weight-related comorbidity (hypertension, type 2 diabetes, and/or dyslipidemia) must be on a stable and allowed treatment regimen for that condition for at least 3 months prior to study enrollment.

6 Participants will be able to provide informed consent before any trial-related activities.

Exclusion Criteria:

1. Women who are pregnant, lactating, or of childbearing potential who are not using adequate contraceptive measures. The following are considered to be adequate methods of birth control: 1.Intrauterine device (IUD); 2. Barrier protection; 3.Contraceptive implantation system (Norplant); 4.Oral contraceptive pills; 5. A surgically sterile partner; and 6. Abstinence. Women who are > 2 years post-menopausal or surgically-sterile are not considered of childbearing potential. All female participants will have a negative pregnancy test prior to randomization.
2. Participants who have made a suicide attempt in the last 10 years, who are displaying clinically significant psychotic features, suicidality, or homicidality on mental status examination, or who have suicidal ideation or behavior as assessed with the C-SSRS.
3. Participants who are receiving behavioral weight loss treatment (BWLT) (e.g., Weight Watchers) that was begun within the 3 months before study entry. Participants who are receiving BWLT that was started 3 months prior to the beginning of the study will be allowed to continue to receive their BWLT during the trial only if they have had no weight loss in the past 3 months and they agree to not make any changes in the frequency or nature of their BWLT during the course of the drug trial.
4. A DSM-5 diagnosis of a substance-related or addictive disorder (except a tobacco-related disorder) within the 3 months prior to enrollment.
5. A DSM-5 diagnosis of dementia, a psychotic disorder, or a depressive disorder.
6. History of any psychiatric disorder which might interfere with a diagnostic assessment, treatment, or compliance.
7. Clinically unstable medical disease, including cardiovascular, hepatic, renal, gastrointestinal, pulmonary, neurological, metabolic, endocrine, or other systemic disease. Clinically stable hypertension, type 2 diabetes, or dyslipidemia are not exclusionary.
8. Have a history of a structural cardiac abnormality, valvular cardiac disease, cardiomyopathy, serious heart rhythm abnormality, coronary artery disease, congestive heart failure, stroke, or other serious cardiovascular problem.
9. Have an ECG with significant arrhythmias or conduction abnormalities, which in the opinion of the physician investigator preclude study participation.
10. Have clinically relevant abnormal laboratory results.
11. Participants requiring treatment with any drug which might interact adversely with or obscure the action of the study medication. This includes anti-obesity drugs, psychostimulants, modafinil or armodafinil, topiramate or zonisamide, and antipsychotics. Participants receiving metformin at a stable dose for ≥ 3 months can be included.
12. Participants receiving GLP-1 based therapies, sodium-glucose co-transporter 2 inhibitors (SGLT2s), thiazolidinediones, sulfonylureas, or insulin.
13. Participants with a personal or family history of medullary thyroid carcinoma or Multiple Endocrine Neoplasia syndrome type 2.
14. Participants who have received any investigational medication within three months prior to randomization.
15. Participants previously screen-failed or randomised to participate in this trial.
16. Participants who have a known or suspected allergy to liraglutide 3.0 mg sc injection, its constituents, or related products.
17. Participants with a urine drug screen positive for a drug that, in the opinion of the investigator, is being abused.
18. Participants with a past medical history of pancreatitis.
19. Participants who had received any investigational drug within 3 months prior to this trial.
20. Participants who require bariatric surgery or are anticipated to require it during the course of the trial. If such surgery becomes warranted during the study, such patients will be excluded from the primary endpoint analysis.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2017-04-26 (Actual); Primary Completion 2022-10-11 (Actual); Study Completion 2023-01-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Lindner Center of HOPE, Mason, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] McElroy SL, Guerdjikova AI, Blom TJ, Mori N, Romo-Nava F. Liraglutide in Obese or Overweight Individuals With Stable Bipolar Disorder. J Clin Psychopharmacol. 2024 Mar-Apr 01;44(2):89-95. doi: 10.1097/JCP.0000000000001803. Epub 2024 Jan 15. PMID 38227621

RESULTS

PARTICIPANT FLOW:
Groups:
- Active Drug: LIRAGLUTIDE 3 Mg/0.5 mL (18 Mg/3 mL) SUB-Q PEN INJECTOR (ML) N=29
- Placebo: Placebo (no active drug) N=31
Period: Overall Study
Arm/Group | Active Drug | Placebo
Started | 29 | 31
Completed | 13 | 8
Not Completed | 16 | 23

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Active Drug | Placebo | Total
Number analyzed (Participants) | 29 | 31 | 60
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 29 | 31 | 60
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.9 (11.0) | 41.4 (12.3) | 42.6 (11.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 24 | 48
  Male | 5 | 7 | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 29 | 31 | 60
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 29 | 31 | 60
Body weight [Mean (Standard Deviation); unit: kg] | 110.6 (24.0) | 101.9 (14.8) | 106.2 (19.1)

OUTCOME MEASURES:

1. Primary Outcome: Percent Change in Body Weight
Description: Percent change in body weight over 40 weeks
Time Frame: 40 week
Population: ≥ 5% of baseline body weight
Measure: Mean (Standard Deviation); unit: % change
Arm/Group | Active Drug | Placebo
Number analyzed (Participants) | 29 | 31
% change | -3.3 (5.2) | 0.2 (4.2)

ADVERSE EVENTS:
Time Frame: Through study completion, for the total duration of the trial, including up to 27 days of screening , the 40 study treatment weeks and one week of follow up
Groups:
- Active Drug: Significantly more placebo recipients (n=11) than liraglutide recipients (n=3) stopped study medication for a side effect (p=0.02). Those who discontinued liraglutide stopped because of gastrointestinal issues (n=1), mood dysregulation (n=1), and suicidal ideation (n=1). No adverse event was judged to reflect an interaction between liraglutide and participants' BD medications. There were no changes in psychopathology safety scales or vital signs. No participants experienced psychosis, displayed suicidal behaviour, or had ECG changes during the study.
- Placebo: Significantly more placebo recipients (n=11) than liraglutide recipients (n=3) stopped study medication for a side effect (p=0.02). Those who discontinued placebo did so for mood dysregulation (n=5), gastrointestinal issues (n=4), and suicidal ideation (n=2). Two participants receiving placebo had a serious adverse event- one was medically hospitalized for a bowel obstruction presumed due to past bariatric surgery while the other was psychiatrically hospitalized for mood dysregulation-neither adverse event was attributed to study medication. There were no changes in psychopathology safety scales or vital signs . No participants experienced psychosis, displayed suicidal behaviour, or had ECG changes during the study.
Arm/Group | Active Drug | Placebo
All-Cause Mortality (participants affected / at risk) | 0/29 | 0/31
Serious Adverse Events (participants affected / at risk) | 0/29 | 2/31
Other Adverse Events (participants affected / at risk) | 29/29 | 25/31
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active Drug (N=29) | Placebo (N=31)
Bowel obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1) — bowel obstruction presumed due to past bariatric surgery
Mood dysregylation (Psychiatric disorders) | 0 (0) | 1 (1) — psychiatric hospitalized for mood dysregulation
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active Drug (N=29) | Placebo (N=31)
Nausea (Gastrointestinal disorders) | 19 (19) | 14 (14)
URI (Respiratory, thoracic and mediastinal disorders) | 10 (10) | 6 (10)
Constipation (Gastrointestinal disorders) | 12 (12) | 3 (3)
Heartburn (Gastrointestinal disorders) | 10 (10) | 2 (2)
Mood dysregulation (Psychiatric disorders) | 7 (7) | 8 (8)
Gastroenteritis (Gastrointestinal disorders) | 7 (7) | 5 (5)
Headache (Nervous system disorders) | 6 (6) | 9 (9)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 7 (7) | 5 (5)
Injection site irritatation (Skin and subcutaneous tissue disorders) | 5 (5) | 6 (6)
Sleep disturbance (Nervous system disorders) | 5 (5) | 5 (5)

LIMITATIONS AND CAVEATS:
The small sample size may have compromised the study's ability to detect important effects. Premature termination rate was high and treatment duration was relatively short. Only individuals with stable BD were enrolled, and therefore results cannot be generalized to individuals with unstable BD.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2017-07-11): https://cdn.clinicaltrials.gov/large-docs/05/NCT03158805/Prot_SAP_000.pdf
  • Informed Consent Form (2018-04-25): https://cdn.clinicaltrials.gov/large-docs/05/NCT03158805/ICF_001.pdf